CLINICAL TRIAL: NCT02443766
Title: Use of a Functional Neuroimaging Battery for the Evaluation of a Meditation
Brief Title: Use of a Functional Neuroimaging Battery for the Evaluation of a Meditation Retreat
Acronym: FETZER
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 11G.488
Record Dates: First submitted 2015-02-06; First posted 2015-05-14 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Integrative Medicine; Alternative Medicine; Complementary Medicine; Meditation Retreat; Ignatian Retreat; Single Photon Emission Computed Tomography (SPECT); Functional Magnetic Resonance Imaging (fMRI); Wellbeing; General Health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Subjects: Healthy subjects will attend the weeklong meditation retreat.
  Interventions: Other: Meditation Retreat

INTERVENTIONS:
Other: Meditation Retreat — Weeklong retreat which includes meditation and prayer.

SUMMARY:
Over 2 decades scientists have been studying the effect on brain function from meditation practices. The purpose of this study is to measure the effect of a meditation retreat program on serotonin and dopamine transporter binding and changes in cerebral blood flow. The retreat program that will be followed is a week-long retreat called the Ignatian Retreat.

DETAILED DESCRIPTION:
This study will utilize DaTscan single photon emission computed tomography (SPECT) and functional magnetic resonance imaging (fMRI) in healthy subjects within one month of entering the retreat. The study uses DaTscan to measure the effect on serotonin and dopamine transporter binding, and functional magnetic resonance imaging (fMRI) to measure the effect on cerebral blood flow. The Ignatian Retreat is a weeklong retreat which involves meditation and prayer.

Additionally, study participants will complete a variety of questionnaires and scales to measure psychological and spirituality states. The scans and questionnaires will be completed before and after the participant has completed the retreat. The ultimate goal of the study is to analyze and compare pre and post imaging and neuropsychological and spirituality changes in healthy controls who participate in this retreat.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent and willing to complete the study.
* Willing to undergo the full imaging procedures.
* Women of childbearing potential with a negative serum pregnancy test.

Exclusion Criteria:

* Any neurological or psychiatric disorders, including drug or alcohol abuse, that may interfere with cerebral blood flow as determined by the principal investigator.
* Any medical conditions that may interfere with cerebral blood flow as determined by the principal investigator.
* Currently taking medication that might affect cerebral blood flow (i.e. antidepressants, antipsychotics, anxiolytics, benzodiazepines, sedatives, antiseizure medications)
* Subject is unable or unwilling to lie still in the scanner (i.e. due to claustrophobia or weight > 350 pounds)
* Subject has metal in their body or other reason that they cannot undergo magnetic resonance imaging.
* Previous brain surgery or intracranial abnormalities they may complicate interpretation of the brain scans. (e.g. stroke, tumor, vascular abnormality).
* Pregnancy
* Allergy to iodine or shellfish.
* Concurrent participation in another research protocol that might affect the outcome of this study as determined by the principle Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At present, study participants are recruited from a variety of meditation programs and through the Center of Integrative Medicine. All subjects will be healthy adults.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Single Photon Emission Computed Tomography (SPECT) Imaging (DaTScan) | Within one month of the retreat
  To detect changes in dopamine and serotonin before and after a meditation retreat program in serotonin transporter and dopamine transporter binding.

SECONDARY OUTCOMES:
functional MRI | Within one month of the retreat
  To detect changes in cerebral blood flow before and after a meditation retreat program.

OTHER OUTCOMES:
Speilberger State Trait Anxiety Inventory (STAI) | Within one month of the retreat
  This validated questionnaire will be used as one of the evaluation questionnaires for the study. The Speilberger State Trait Anxiety Inventory (STAI) contains a total of 40 questions, half of which relate to the way subjects are feeling at the moment and half of which ask them to describe how they usually feel.
Profile of Moods Scale (POMS) | Within one month of the retreat
  The Profile of Mood States (POMS) is a validated questionnaire of 65 single word items that asks "How have you been feeling in the past week including today." The subjects will select their response to each word that describes a mood or feeling on a Likert scale from 1= Not at All, 2= A Little, 3=Moderately, 4=Quite a lot, to 5=Extremely. The responses are scored to generate values for Tension, Anger, Confusion, Depression and Vigor. The higher scores indicate a greater presence of that mood or state.
Beck Depression Inventory (Beck 1972) | Within one month of the retreat
  This validated questionnaire will be used as one of the evaluation questionnaires for the study. The Beck Depression Inventory (Beck 1972) is a standard 21 item questionnaire probing cognitive and somatic symptoms of depression. The higher scores indicate a greater presence of depression.
Standard Form-12 (SF-12) | Within one month of the retreat
  This 12-item validated questionnaire will be used as one of the evaluation questionnaires for the study. The subjects will select their response to each word that describes a mood or feeling on a Likert scale.
Hood Mysticism Scale (Lifetime) | Within one month of the retreat
  This validated scale will be used as one of the evaluation questionnaires for the study. Items are rated on a five-point scale with negatively worded items reverse scored. The responses are scored to generate values for Extrovertive Mysticism, Religious Interpretation, and Introvertive Mysticism.
Brief Multidimensional Measure of Religiousness/Spirituality | Within one month of the retreat
  This 30-item validated questionnaire will be used as one of the evaluation questionnaires for the study. The responses are scored to generate values for Suffering, Positing Sharing, Crying, Emotional Attention, Feel for Others, and Emotional Contagion.
Gratitude Questionnaire | Within one month of the retreat
  This validated questionnaire will be used as one of the evaluation questionnaires for the study. The subjects will select their response on a Likert scale. The higher scores indicate a greater sense of gratitude.
Daily Spiritual Experience Scale | Within one month of the retreat
  This validated questionnaire will be used as one of the evaluation questionnaires for the study. This assessment measures ordinary, or daily, spiritual experiences.
The Assessment of Spirituality and Religious Sentiments (ASPIRES ) | Within one month of the retreat
  This validated questionnaire will be used as one of the evaluation questionnaires for the study. This assessment measures Religious sentiments and Spiritual Transcendence.
Index of Core Spiritual Experiences (INSPIRIT) | Within one month of the retreat
  This validated questionnaire will be used as one of the evaluation questionnaires for the study to evaluate the presence or frequency of certain religions.
Functional Assessment of Chronic Illness Therapy Spiritual Well-Being (FACIT-Sp-12) | Within one month of the retreat
  This validated questionnaire will be used as one of the evaluation questionnaires for the study. The 12-item assessment is used to measure spiritual well-being by asking patients to describe aspects of spirituality and/or religious faith that contribute to health related quality of life.
Cloninger Self-Transcendence Scale | Within one month of the retreat
  This validated questionnaire will be used as one of the evaluation questionnaires for the study. The subjects will select their response on a Likert scale. The higher scores indicate a greater presence to self-transcendence and well being.
Five Facet Mindfulness Questionnaire | Within one month of the retreat
  This validated questionnaire will be used as one of the evaluation questionnaires for the study.The analysis yielded five factors that appear to represent elements of mindfulness as it is currently conceptualized.The five facets are observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B. Newberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Publication from study results — http://www.andrewnewberg.com/journal-articles/effect-of-a-one-week-spiritual-retreat-on-dopamine-and-serotonin-transporter-binding-pdf-a-preliminary-study

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-12-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT02443766/Prot_SAP_002.pdf